CLINICAL TRIAL: NCT05942170
Title: The Combination of Preoperative MRI and Sentinel Lymph Node Biopsy（SLN） in the Surgical Management of Cervical and Endometrial Cancer
Brief Title: The Combination of Preoperative MRI and SLN in the Surgical Management of CC and EC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAHoWMU-CR2023-07-101
Record Dates: First submitted 2023-02-19; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-02

CONDITIONS: Sentinel Lymph Node Biopsy; MRI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SLN/MRI (Other)
  Interventions: Drug: ICG/ blue dye

INTERVENTIONS:
Drug: ICG/ blue dye — The SLN mapping procedure was performed as previously described by using IGC or blue dye. The injection technique of the tracers was the same for both cervical and endometrial cancer. The cervical injection was done by insulin syringe(one ml) inserting full needle length (1 cm) and complete injection at 3, 9 o'clock, or 2,4,8,10 o'clock.

SUMMARY:
The aim of the study was to evaluate the diagnostic value of MRI and/or SLN mapping alone or in combination in cervical (CC) and endometrial cancer (EC) patients.

DETAILED DESCRIPTION:
Cervical (CC) and endometrial cancer (EC) are the most common female malignancies after breast cancer. Cervical cancer is one of the three primary malignant tumors of the female reproductive system. According to the 2018 global cancer statistics, Cervical cancer is the 4th most common cancer among women. According to 2020 data there were 16,607 fatal cases and 81,964 new cases of endometrial cancer in China. The presence of pelvic lymph node metastases is the primary poor prognostic marker in the early stages, and the state of para-aortical lymph nodes is an essential predictor of relapse. Compared with patients without lymph node metastasis which get 90-95% five-year survival rates, the patients with pelvic and para-aortic metastatic lymph nodes were only in 50% and 20-30%, respectively.

On the one hand, A previous study reported that pelvic lymph node metastasis was detected in less than 5% of patients with stage IA endometrial cancer but more than 90% of patients with early-stage endometrial cancer underwent unnecessary comprehensive pelvic lymphadenectomy. On the other hand, Lymph nodal status represents a crucial piece of information for the oncologic management of cervical cancer patients. Surgical and pathological diagnosis of lymph nodes is the gold standard for identifying tumor stage of CC and high-risk EC. When lymph nodes metastasis are existed in EC or CC, the treatment approaches may change. A hysterectomy without lymphadenectomy is advised in stage IA1 CC without lymphovascular invasion. It is advised to add a pelvic lymphadenectomy in stages IA2-IB1,and additional adjuvant treatment is recommended once lymph node metastasis is confirmed. The Clinical guidelines of the therapy for high-risk EC is bilateral adnexectomy and radical hysterectomy.Endometrial cancer surgical treatment still remains controversial, particularly when the disease is in its early stages. According to the study, individuals with early-stage endometrial cancer may not receive any therapeutic benefit from a full lymphadenectomy.

However, comprehensive lymphadenectomy has many serious complications including lower extremity lymphedema, pelvic lymphocele, significant bleeding, nerve damage, and postoperative ileus etc. Comprehensive lymphadenectomy may compromise specific healthy lymph nodes' barrier and immunological functions, even to the extent that raising the chance of undetected cancer foci distant metastasizing. Inflammation, tumor size, malignant emboli, compression, physician detection approach, and patient history of neoadjuvant chemotherapy all impact the detection rate and Sensitivity of SLN.

The SLN mapping must have a small proportion of false-negative findings to be considered credible. To put it another way, a pathologically negative SLN must accurately reflect a pathologically negative condition of the ipsilateral pelvis. However, several prospective investigations show that the techniques have weak Sensitivity and a low positive predictive value below a generally recognized criterion of 90%.In this case, a non-invasive strategy has been applied to evaluate the occurrence of lymph node metastases using several imaging modalities. Magnetic resonance imaging (MRI) is the imaging modality used in the initial work-up to study the primary tumor and pelvic lymph node involvement. The use of imaging technologies, such as CT, MRI, PET, and DWI, may enable the accurate detection of pelvic and para-aortic LN metastases in cervical cancer patients as medical science and technology advance. Based on assessments of node size and/or morphologic information, LN metastases have traditionally and widely been detected using MRI.

Aiming to detect early CC and EC patients with lymph node metastases, our study evaluated the Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the preoperative MRI and SLN mapping, alone or in combination, try to find a simpler and safer method for correct diagnosis of lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* histopathological diagnosis of cervical cancer or endometrial cancer
* complete case data
* preoperative MRI examinations completed
* initial treatment is surgical
* all surgeries are entirely staged.

Exclusion Criteria:

* patients with suspected extrauterine involvement
* allergic to tracers
* previous history of surgery or radiotherapy to nodal areas
* contraindication for surgical treatment (due to age or comorbidities).

Ages: 41 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the preoperative MRI and SLN mapping, alone or in combination | 7 days
  Clinical-pathologic characteristics were evaluated using basic descriptive statistics. The Sensitivity, of MRI, SLN biopsy, and the combination of MRI and SLN biopsy in identifying metastatic lymph nodes were calculated. A true positive was defined as a positive MRI or SLN in the presence of metastatic disease to the pelvic lymph nodes. A true negative was defined as a negative MRI and SLN in the absence of metastatic disease to the pelvic lymph nodes. A false positive was defined as a positive MRI in the absence of metastatic disease to the pelvic lymph nodes. A false negative was defined as a negative MRI or SLN in the presence of metastatic disease in the pelvic lymph nodes. Ninety-five percent confidence intervals (CIs) were calculated according to the standard normal distribution. These analyses were performed for the entire population. Statistical analysis was performed with GraphPad Prism 9.
specificity of the preoperative MRI and SLN mapping, alone or in combination | 7 days
  Clinical-pathologic characteristics were evaluated using basic descriptive statistics. The specificity, of MRI, SLN biopsy, and the combination of MRI and SLN biopsy in identifying metastatic lymph nodes were calculated. A true positive was defined as a positive MRI or SLN in the presence of metastatic disease to the pelvic lymph nodes. A true negative was defined as a negative MRI and SLN in the absence of metastatic disease to the pelvic lymph nodes. A false positive was defined as a positive MRI in the absence of metastatic disease to the pelvic lymph nodes. A false negative was defined as a negative MRI or SLN in the presence of metastatic disease in the pelvic lymph nodes. Ninety-five percent confidence intervals (CIs) were calculated according to the standard normal distribution. These analyses were performed for the entire population. Statistical analysis was performed with GraphPad Prism 9.
positive predictive value (PPV) of the preoperative MRI and SLN mapping, alone or in combination | 7 days
  Clinical-pathologic characteristics were evaluated using basic descriptive statistics. The PPV of MRI, SLN biopsy, and the combination of MRI and SLN biopsy in identifying metastatic lymph nodes were calculated. A true positive was defined as a positive MRI or SLN in the presence of metastatic disease to the pelvic lymph nodes. A true negative was defined as a negative MRI and SLN in the absence of metastatic disease to the pelvic lymph nodes. A false positive was defined as a positive MRI in the absence of metastatic disease to the pelvic lymph nodes. A false negative was defined as a negative MRI or SLN in the presence of metastatic disease in the pelvic lymph nodes. Ninety-five percent confidence intervals (CIs) were calculated according to the standard normal distribution. These analyses were performed for the entire population. Statistical analysis was performed with GraphPad Prism 9.
negative predictive value (NPV) of the preoperative MRI and SLN mapping, alone or in combination | 7 days
  Clinical-pathologic characteristics were evaluated using basic descriptive statistics. The NPV of MRI, SLN biopsy, and the combination of MRI and SLN biopsy in identifying metastatic lymph nodes were calculated. A true positive was defined as a positive MRI or SLN in the presence of metastatic disease to the pelvic lymph nodes. A true negative was defined as a negative MRI and SLN in the absence of metastatic disease to the pelvic lymph nodes. A false positive was defined as a positive MRI in the absence of metastatic disease to the pelvic lymph nodes. A false negative was defined as a negative MRI or SLN in the presence of metastatic disease in the pelvic lymph nodes. Ninety-five percent confidence intervals (CIs) were calculated according to the standard normal distribution. These analyses were performed for the entire population. Statistical analysis was performed with GraphPad Prism 9.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhao, master, Study Chair — The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU
Locations (1):
- The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang, China